CLINICAL TRIAL: NCT07200622
Title: Evaluating the Effects of GLP-1 Analogue, Oral Semaglutide, in Patients With Alzheimer's Disease
Brief Title: Oral Semaglutide in Patients With Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21HH7080
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: GLP-1 Analogues; Semaglutide; Alzheimers
MeSH Terms: conditions — Alzheimer Disease | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: A 12-month, multicentre, randomised, double-blind, placebocontrolled study in patients with mild to moderate Alzheimer's dementia. Subjects will be randomised on a 1:1 ratio to receive oral semaglutide or matching placebo. Participants will be maintained at the highest well-tolerated daily dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Rybelsus) (Experimental)
  Interventions: Drug: Semaglutide (Rybelsus®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) — All subjects will receive oral semaglutide once daily (4-weekly dose escalation from 3 mg to 7 mg and finally 14 mg). This dose escalation schedule is specified in the IMP (Rybelsus) SmPC.
  Arms: Semaglutide (Rybelsus)
Drug: Placebo — Matched oral Placebo to be taken once daily.
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is a progressive neurodegenerative disease and a major global healthcare burden. Currently, the disease is only treated symptomatically and an effective disease-modifying therapy (DMT) that may slow the disease progression, and prevent cognitive and functional deterioration, is yet to emerge. Glucagon-like peptide-1 (GLP-1) analogues are being studied to treat neurodegenerative diseases, due to evidence of their neuroprotective effects in mouse models of AD. This study investigates Semaglutide, a modified human GLP-1RA in Alzheimer's disease to understand the mechanism of the disease. The primary objective of this study is to evaluate the safety and tolerability of oral semaglutide in individuals with mild AD. Moreover, the secondary objective of the study is to evaluate the change in synaptic density using PET before and after treatment with semaglutide.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving and capacity to give informed consent.
2. An individual who can act as a reliable study partner with regular contact
3. Diagnosis of Alzheimer's disease according to the revised NIA-AA criteria
4. Age from 50 years
5. Mini-Mental State Examination (MMSE) score of ≥18; likely complete all the assessments
6. Rosen Modified Hachinski Ischemic score ≤4
7. On stable medication for 2 months before the screening visit; on or off cholinesterase inhibitors
8. Fluency in English and evidence of adequate premorbid intellectual functioning
9. Likely to be able to participate in all scheduled evaluations and complete all required tests

Exclusion Criteria:

1. Any contraindications to the use of oral semaglutide
2. Significant neurological disease other than AD that may affect cognition
3. MRI/CT showing unambiguous aetiological evidence of cerebrovascular disease with regard to their dementia or vascular dementia fulfilling NINCDSAIREN criteria
4. Current presence of a clinically significant major psychiatric disorder
5. Current clinically significant systemic illness that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study
6. Myocardial infarction within the last 1 year
7. Other clinically significant abnormality on physical, neurological or laboratory examination that could compromise the study or be detrimental to the subject
8. History of alcohol or drug dependence within the last 2 years
9. Current use of narcotic medications which could affect cognition. Subjects on anticoagulants will be allowed, but will not have an arterial line inserted
10. Women of childbearing potential. Women who could become pregnant will be required to use adequate contraception throughout the trial. Please see appendix A for more information. All women of childbearing potential will take a pregnancy test before the PET scan.
11. Any contraindications to MRI scanning
12. Any historical evidence of pancreatitis or gallstones as proven by ultrasound or medical admission.
13. History of medullary thyroid cancer
14. Patients diagnosed with T2DM who are unwilling to change their treatment to semaglutide.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of oral semaglutide in an AD population. | Adverse events monitoring: Baseline; Weeks 4, 8, 26, 39, 52
  To assess the safety and tolerability of (1-year) Semaglutide treatment in patients with AD using composite outcome measure of the adverse events evaluated from the safety assessments. This will be assessed by the number of participants using a composite measure generated from abnormal vital signs, abnormal 12-lead ECG readings, abnormal laboratory (blood) tests, abnormalities found in MRI scans, abnormal physical exam findings, and abnormal neurological/psychiatric evaluation.

SECONDARY OUTCOMES:
To evaluate the change in synaptic density using [18F] SynVesT-1 before and after treatment. | [18F] SynVesT-1 PET will be conducted at baseline and Week 52 (end of treatment).
  Synaptic density will be assessed, using [18F] SynVesT-1, at baseline and after 1-year of treatment with Semaglutide.

IPD SHARING:
Plan to Share IPD: Undecided